CLINICAL TRIAL: NCT02799459
Title: Evaluation of Medical and Economic Incidence of Hypnosis in Conization
Brief Title: Evaluation of Medical and Economic Incidence of Hypnosis
Acronym: HYPNONISAT°
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Mutualiste de Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 15-MUTG-01
Record Dates: First submitted 2016-06-03; First posted 2016-06-14 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Surgery
Keywords: Hypnoanesthesia; Hypnosis; conization
MeSH Terms: interventions — Anesthesia, General; Hypnosis; Conization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- General anaesthesia: this group will allow us to compare the results like it is the treatment used in current practice ie general anesthesia.
  Interventions: Procedure: General anaesthesia
- Hypnosis in conization: This group is the treatment being tested , where hypnosis is used in the conization
  Interventions: Procedure: Hypnosis in conization

INTERVENTIONS:
Procedure: General anaesthesia — the patient will receive a general anaesthesia do proceed at her conization
  Groups: General anaesthesia
Procedure: Hypnosis in conization — this is the experimental treatment which is allocated to the experimental group
  Groups: Hypnosis in conization

SUMMARY:
Hypnosis in conization is more and more use to substitute General Anesthesia (GA) in Anesthesia's field.

This study wants to prove that the Hypnosis in conization are cheaper.

DETAILED DESCRIPTION:
Hypnosis in conization is more and more use to substitute General Anesthesia (GA) in Anesthesia's field. There are few studies about this new anesthesia tool. The latter showed that it's possible to substitute GA by hypnosis. This tool could have many positive such as reduced pains, anxiety or post operative vomiting nausea (POVN). Hypnosis in conization also allows time reduction in post operative security monitoring room (SSPI), speedier hospital discharge and greater patient satisfaction. Most studies involves 1 or 2 practitioners and few patients. There is no reliable research which compare Hypnosis in conization costs and GA costs. Since 2010, anesthesia's team of Grenoble Mutualist Hospital group (GHM) realized many Hypnosis in conization surgical procedures. Half of the team had been trained to Hypnosis in conization and use it for several types of surgeries for a lot of surgeons. It's the case for conisations. Currently, the 7 gynaecologists surgeons of the team achieved between 150 and 200 per year , some of this used GA, others used Hypnosis in conization, and unusually they used " rachianesthesia ". Thus, it gives us the opportunity for studying Hypnosis in conization, without practitioner effect, for a relatively cohesive group of patients (vast majority of patients are between 30 and 50 years and they haven't any particular medical history).

ELIGIBILITY:
Inclusion Criteria:

* all women whom need a conization

Exclusion Criteria:

* age<18 ans
* guardianship
* trusteeship
* not affiliated to the social security

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all women whom need a conization
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
economic benefit of Hypnosis in conization compare to GA | 1 month
  The primary study endpoint will be the GA costs compare to Hypnosis in conization costs

SECONDARY OUTCOMES:
time spent in the operating room | 1 day
time spent in SSPI | 1 day
time of participation in out-patient surgery department | 1 day
hospital admission rates | 1 year
postoperative pain using a visual analog scale | up to 1 month
time to resumption of professional activity | 3 months
patients satisfaction using a visual analog scale | up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jerome Schweitzer, Physician, Principal Investigator — Groupe Hospitalier Mutualiste de Grenoble
Locations (1):
- Groupe Hospitalier Mutualiste de Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Defechereux T, Faymonville ME, Joris J, Hamoir E, Moscato A, Meurisse M. [Surgery under hypnosedation. A new therapeutic approach to hyperparathyroidism]. Ann Chir. 1998;52(5):439-43. French. PMID 9752483
- [Background] Sefiani T, Uscain M, Sany JL, Grousseau D, Marchand P, Villate D, Vincent JL. [Laparoscopy under local anaesthesia and hypnoanaesthesia about 35 cholecystectomies and 15 inguinal hernia repair]. Ann Fr Anesth Reanim. 2004 Nov;23(11):1093-101. doi: 10.1016/j.annfar.2004.08.014. French. PMID 15581727
- [Background] Defechereux T, Degauque C, Fumal I, Faymonville ME, Joris J, Hamoir E, Meurisse M. [[Hypnosedation, a new method of anesthesia for cervical endocrine surgery. Prospective randomized study]. Ann Chir. 2000 Jul;125(6):539-46. doi: 10.1016/s0003-3944(00)00238-8. French. PMID 10986765
- [Background] Faymonville EM, Mambourg HP, Joris J, Vrijens B, Fissette J, Albert A, Lamy M. Psychological approaches during conscious sedation. Hypnosis versus stress reducing strategies: a prospective randomized study. Pain. 1997 Dec;73(3):361-367. doi: 10.1016/S0304-3959(97)00122-X. PMID 9469526